CLINICAL TRIAL: NCT03899129
Title: Effect Of Simultaneous Working Length Control During Root Canal Preparation Versus Electronic Apex Locator On Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis (a Randomized Clinical Trial)
Brief Title: Effect Of Simultaneous Working Length Control Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aml mohammed Abdel moteleb, master degree student, Endodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2019-03-02
Record Dates: First submitted 2019-03-08; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Type: Two arm, parallel, randomized clinical trial. Allocation ratio: 1:1 Framework: Superiority.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be participant-blind where the participants will not know the intervention done. The applications could not be blinded; however, the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simultaneous working length control (Experimental): • Using simultaneous working length control during root canal preparation using E-CONNECT S endomotor with integrated apex locator.
  Interventions: Procedure: simultaneous working length control using E-CONNECT S
- Root ZX apex locator. (Active Comparator): Using manual control of the working length by using stoppers during instrumentation (separate length determination and root canal preparation) using Root ZX apex locator.
  Interventions: Procedure: separate length determination and root canal preparation using Root ZX apex locator.

INTERVENTIONS:
Procedure: simultaneous working length control using E-CONNECT S — E-CONNECT S (Eighteeth medical technology Co., Ltd, china) is an endomotor with integrated apex locator newly introduced in the market with continuous WL measuring function. It contains an optional module for rotary instrumentation, allowing the device to function as a low-speed handpiece, apex locator, or a combination of both. This motor has an attention-grabbing property that when an instrument reaches the predetermined working length, the motor automatically stops the instrumentation. Thus, it can be concluded that automatically stopping instrumentation when the instrument reaches the working length would decrease postoperative pain compared with manually controlling the working length by using stoppers during instrumentation (separate length determination and root canal preparation).
  Arms: simultaneous working length control
Procedure: separate length determination and root canal preparation using Root ZX apex locator. — Using manual control of the working length by using stoppers during instrumentation (separate length determination and root canal preparation) using Root ZX apex locator.
  Arms: Root ZX apex locator.

SUMMARY:
The aim of this study was to evaluate the effect of simultaneous length control during root canal preparation on postoperative pain compared with separate working length determination and root canal preparation using electronic apex locator. During preparation of root canals, loss of working length (WL) can lead to instrumentation beyond the predefined apical limit of the preparation. This effect is mainly attributed to straightening of the root canal during instrumentation. Some studies showed, that this kind of over instrumentation as well as under instrumentation can adversely affect the outcome of the endodontic treatment, while it remains uncertain what exactly is the most favorable extent of the apical limit of root canal preparation. Furthermore, all endodontic instruments produce apical extrusion of debris, even when the preparation is kept within the confines of the root canal. Consequently, preparations ending in the periapical tissue will produce a greater amount of debris extrusion that could elicit a neurogenic inflammatory response resulting from an irritation of the periodontal ligament with subsequent postoperative symptomatic apical periodontitis. Therefore, it seems favorable to control the determined WL during root canal preparation to avoid preparations ending in the periapical tissue.

DETAILED DESCRIPTION:
During preparation of root canals, loss of working length (WL) can lead to instrumentation beyond the predefined apical limit of the preparation. This effect is mainly attributed to straightening of the root canal during instrumentation. Some studies showed, that this kind of over instrumentation as well as under instrumentation can adversely affect the outcome of the endodontic treatment. Furthermore, all endodontic instruments produce apical extrusion of debris, even when the preparation is kept within the confines of the root canal. Consequently, preparations ending in the periapical tissue will produce a greater amount of debris extrusion that could result from an irritation of the periodontal ligament with subsequent postoperative symptomatic apical periodontitis. Therefore, it seems favorable to control the determined WL during root canal preparation to avoid preparations ending in the periapical tissue.

Endodontic motors with integrated apex locators offer a solution to the described problem as they have been developed with the intention of making root canal treatment easier and faster. Besides torque and speed control, these devices also aim to continuously monitor and control the apical limit all the way through the mechanical preparation of the root canals and have an auto apical reverse (AAR) function that stops and reverse the rotation when the file tip reaches the predetermined apical limit of the preparation.

E-CONNECT S (Eighteeth medical technology Co., Ltd, china) is an endomotor with integrated apex locator newly introduced in the market with continuous WL measuring function. It contains an optional module for rotary instrumentation, allowing the device to function as a low-speed hand piece, apex locator, or a combination of both. This motor has an attention-grabbing property that when an instrument reaches the predetermined working length, the motor automatically stops the instrumentation. Thus, it can be concluded that automatically stopping instrumentation when the instrument reaches the working length would decrease postoperative pain compared with manually controlling the working length by using stoppers during instrumentation (separate length determination and root canal preparation).

The Root ZX (J Morita, Tokyo, Japan) is a third generation EAL where no calibration is necessitated, and a microprocessor analyzes the impedance quotient. It uses multiple frequencies to calculate the distance from the end of the canal. To measure location within the canal, third generation units (including Root ZX EAL) still use impedance measurements but have stronger microprocessors and can process the mathematical quotient and algorithm calculations required to obtain accurate readings. The change in electrical capacitance at the apical constriction is the basis for the operation of the Root ZX and its reported accuracy, even in presence of different electrolytes in the canal and under different clinical conditions; that's why it is considered the most commonly used apex locator.

ELIGIBILITY:
Inclusion Criteria:

* Age between (20-50) years old with symptomatic irreversible pulpitis in permanent mandibular premolar teeth.
* Systemically- healthy patients (ASA I or II).
* Patients who agree to attend for recall appointments and provide written consent.

Exclusion Criteria:

* Pregnant women and patients with pacemakers.
* Patients with bruxism or clenching or have taken analgesics during past 24 hours.
* Moderate or severe marginal periodontitis (i.e. pocket probing >3 mm).
* Necrotic pulp, pulp polyp, tooth tender to percussion, preoperative palpation pain, clinical progression into periapical abscess, fistula.
* Teeth with internal or external resorption, curvatures, open apices, root canal obliteration, perforation, incomplete root formation, teeth previously undergone root canal treatment, absence of opposing tooth to the related tooth or radiographically invisible canals.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain after endodontic treatment | 7 days after root canal treatment.
  Intensity of postoperative pain will be measured using Visual Analogue scale (VAS) for pain assessment 7 days after the end of endodontic treatment. It uses numerical data:
  None 0, Mild <20, Moderate 20-50 and Sever >50.

SECONDARY OUTCOMES:
Number of analgesic tablets taken by the patient after endodontic treatment. | Until 7 days after endodontic treatment.
  Number of analgesic tablets taken by the patient after endodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aml M moteleb, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 6 months from study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.